CLINICAL TRIAL: NCT00688727
Title: Cognitive Behavioural Therapy in Dissociative Seizures: A Randomised Controlled Trial
Brief Title: Cognitive Behavioural Therapy in Dissociative Seizures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Collaborators: Special Trustees for St Thomas' and Guy's Hospitals (Unknown)
Responsible Party: Dr John Mellers, South London and Maudsley NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R000726
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Dissociative Seizures
Keywords: non epileptic seizures; cognitive behavioural therapy; dissociative disorders; Seizure disorders; randomised controlled trial
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Seizures; Dissociative Disorders; Epilepsy | interventions — Cognitive Behavioral Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive behavioural Therapy
  Interventions: Behavioral: CBT
- 2 (Active Comparator): Standard Care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: CBT — CBT, up to 12 sessions.
  Other Names: Cognitive Behavioural Therapy
  Arms: 1
Behavioral: Standard Care — Routine review by neuropsychiatrist in outpatient clinic
  Other Names: Standard medical care
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether adults with disoociative (psychogenic non-epileptic) seizures receiving cognitive behavioural therapy (CBT) show a greater reduction in seizures and health service use and greater improvement in employment status and overall psychosocial functioning than patients who receive standard care.

DETAILED DESCRIPTION:
Preliminary results from a pilot study demonstrated that cognitive behavioural therapy (CBT) is associated with a significant benefit for patients with dissociative seizures. The current study aims to extend these findings by conducting a randomised controlled trial comparing CBT with standard outpatient medical care. Standard outpatient care has been chosen as the comparison treatment as it most closely resembles what is currently offered to this group of patients by the National Health Service. The primary outcome measure will be seizure frequency. Secondary outcome measures will be work and social adjustment and health service use.

Our hypothesis is that CBT will be superior to standard outpatient care for patients with dissociative seizures as determined by the above measures.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of dissociative seizures
* diagnosis confirmed by video EEG telemetry where practicable
* aged 16 - 70

Exclusion Criteria:

* co existent diagnosis (past or present) of epilepsy
* seizure frequency of less than 2 seizures per month
* current alcohol or drug abuse
* benzodiazepine use exceeding the equivalent of 10mg diazepam per day.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2001-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
seizure frequency | previous month

SECONDARY OUTCOMES:
seizure freedom | 3 months
Work & Social Adjustment scale (Marks, 1986) | Pre-treatment, end of treatment and six-months follow-up
Employment Status | Pre-treatment, end of treatment and six-months follow-up
Health Service Use | Pre-treatment, end of treatment and six-months follow-up
Hospital Anxiety and Depression Scale (Zigmond & Snaith, 1983) | Pre-treatment, end of treatment and six-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goldstein, Study Director — Institute of Psychiatry; John Mellers, Principal Investigator — Maudsley Hospital
Locations (1):
- Maudsley Hospital, London, United Kingdom

REFERENCES:
- [Background] Goldstein LH, Deale AC, Mitchell-O'Malley SJ, Toone BK, Mellers JD. An evaluation of cognitive behavioral therapy as a treatment for dissociative seizures: a pilot study. Cogn Behav Neurol. 2004 Mar;17(1):41-9. doi: 10.1097/00146965-200403000-00005. PMID 15209224